CLINICAL TRIAL: NCT03394937
Title: Study to Assess the Safety and Tolerability of ECI-006 mRNA Immunotherapy by Intranodal Administration in Melanoma: (1) Following Surgical Resection, and (2) in Patients With Stable Disease After Standard of Care Immunotherapy Treatment
Brief Title: Safety of Intranodal ECI-006 in Melanoma Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Expiry of study medication
Sponsor: eTheRNA immunotherapies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E011-MEL
Record Dates: First submitted 2017-11-28; First posted 2018-01-09 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2020-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: • Drug: ECI-006 mRNA Cohort 1: 5 intranodal injections of either 600 µg or 1800 µg mRNA Cohort 2: 9 intranodal injections of either 1800 µg or 3600 µg mRNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 600 µg ECI-006 (Experimental): Patients with melanoma are planned to be dosed intranodal with up to 5 doses of 600 µg ECI-006
  Interventions: Biological: ECI-006
- Cohort 1 1800 µg ECI-006 (Experimental): Patients with melanoma are planned to be dosed intranodal with up to 5 doses of 1800 µg ECI-006
  Interventions: Biological: ECI-006
- Cohort 2 1800 µg ECI-006 (Experimental): Patients with melanoma are planned to be dosed intranodal with up to 9 doses of 1800 µg ECI-006
  Interventions: Biological: ECI-006
- Cohort 2 3600 µg ECI-006 (Experimental): Patients with melanoma are planned to be dosed intranodal with up to 9 doses of 3600 µg ECI-006
  Interventions: Biological: ECI-006

INTERVENTIONS:
Biological: ECI-006 — ECI-006 consists of TriMix and 5 tumor associated antigens mRNA. TriMix is a mixture of mRNAs that encodes potent immune stimulating molecules

SUMMARY:
The purpose of this study is to assess the safety and tolerability of cancer immunotherapy ECI-006 and to determine its ability to induce a measurable immune response against the tumor associated antigens.

In Cohort 1, ECI-006 will be administered 5 times by intranodal injection in melanoma patients after resection of their tumor.

In Cohort 2, ECI-006 will be administered 9 times by intranodal injection on top of standard of care anti PD1 in metastatic melanoma patients with stable disease after 3 to 12 months treatment.

ECI-006 activates key immunologically active cells to direct the immune system against the cancer. Expected potential risks for ECI-006 are non-serious and related to the local administration of the product. Hence, the therapy suggested here has the promise to offer considerable benefit to patients without any major risk.

ELIGIBILITY:
Main inclusion criteria Cohort 1:

1. Age greater than or equal to 18 years and less than or equal to 80 years.
2. Patients must have histologically proven primary malignant melanoma of skin which has been surgically removed (see exclusion criterion on patients with primary uveal melanoma or melanoma of the mucosae).
3. Patients with American Joint Committee on Cancer (AJCC) Stage IIc, III or IV.
4. Patients must have no evidence of disease as evidenced by a whole body 18F fluorodeoxyglucose (FDG) positron emission tomography [PET]/computed tomography [CT] scan to be done at maximum 2 weeks before Visit 2. To exclude the presence of tumor lesions in the brain magnetic resonance imaging (MRI) may be performed.
5. Full recovery from all prior therapies. A maximum period of 12 weeks following major surgery, or any other major invasive procedure is allowed before start of the study medication; at least 4 weeks should be between major surgery and the start of the immunotherapy
6. Female patients of childbearing potential should have a negative serum pregnancy test at Visit 1 (Screening) and should use an efficient method of birth control from screening until the first menses after a 4 week period after the last dose of study medication.

Main exclusion criteria Cohort 1:

1. Patients with primary uveal or mucosal melanoma.
2. Patients who have received prior systemic therapy and/or active immunotherapy for melanoma, such as antigen loaded dendritic cells or chimeric antigen receptor (CAR) T cells, are excluded. Systemic adjuvant treatment for melanoma that is more than 5 years ago and prior local treatment of primary and metastatic tumor lesions (e.g., surgical resection, isolated limb perfusion radiotherapy) are allowed.
3. Patients with a history of autoimmune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, rheumatoid arthritis or multiple sclerosis. Vitiligo is not an exclusion criterion
4. Patients with serious intercurrent chronic or acute illness such as pulmonary [asthma or chronic obstructive pulmonary disease (COPD)] or cardiac (New York Heart Association [NYHA] class III or IV) or hepatic disease or other illness considered by the investigator to constitute an unwarranted high risk for investigational drug treatment.
5. Concurrent second malignancy other than non-melanoma skin cancer, or controlled superficial bladder cancer. In the event of prior malignancies treated surgically, the patient must be considered NED (no evidence of disease) for a minimum of 3 years prior to enrolment.
6. Patients on steroid therapy > 10 mg prednisone (or equivalent) or other immunosuppressive agents such as azathioprine or cyclosporine A (but not limited to these) are excluded on the basis of potential immune suppression. Patients must have had 8 weeks of discontinuation of any steroid therapy exceeding > 10 mg prednisone (or equivalent) before first dose.

Main inclusion criteria Cohort 2:

1. Histologically confirmed AJCC Stage III or Stage IV unresectable disease.
2. Patient must be free of progression and have stable disease after at least 3 months but less than 12 months of first-line immunotherapy (pembrolizumab, nivolumab or combination of nivolumab and ipilimumab). Patients with clinically stable disease can be either:

   1. Patients with stable disease as defined by RECIST1.1 criteria as assessed on 2 consecutive imagings, or
   2. Patients deemed unlikely to respond further to the standard of care immunotherapy by the investigator, after an initial partial response.
3. Patient must continue with standard of care pembrolizumab or nivolumab during the study.
4. Measurable disease by means of clinical examination, computed tomography (CT) or magnetic resonance imaging (MRI) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, defined as:

   * At least 1 tumor lesion that can be accurately and serially measured in at least 1 dimension, and for which the greatest diameter is ≥ 10 mm or at least one malignant lymph node for which the short axis is ≥ 15 mm as measured by contrast enhanced or spiral CT scan and/or
   * At least 1 superficial cutaneous melanoma lesion ≥ 10 mm as measured by calipers and/or
   * At least 1 subcutaneous melanoma ≥ 10 mm lesion and/or
   * Multiple superficial melanoma lesions which in aggregate have a total diameter of ≥ 10 mm

Main exclusion criteria Cohort 2:

1. Patient who received radiotherapy within 4 weeks prior to the start of treatment with study medication.
2. Patients with active brain metastases. Patients with brain metastases are eligible if the brain metastases are deemed stable and if the patient is eligible to receive pembrolizumab as standard of care to treat his melanoma in the judgement of the investigator. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 8 weeks prior to study drug administration.
3. Patients with primary uveal or mucosal melanoma.
4. Patients that are deemed at risk for autoimmune flare up (e.g. patients that had an ongoing/recurrent irAE in the last 3 months), as determined by the investigator.
5. Patients who have received prior treatment for advanced melanoma other than standard of care first-line immunotherapy (pembrolizumab, nivolumab or nivolumab/ipilimumab combination) and targeted therapy (encorafenib, dabrafenib and trametinib) for BRAF positive patients preceding standard of care immunotherapy..

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs), including the incidence of dose-limiting toxicities (DLTs), graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | 24 weeks
  Types of toxicities, incidences and severity will be summarized by descriptive statistics

SECONDARY OUTCOMES:
Immune response associated with ECI-006 administration | 24 weeks
  Antigen-specific T cell responses will be investigated at several time points

CONTACTS AND LOCATIONS:
Locations (9):
- Belgium (5):
  - 032-004_GZA Sint-Augustinus, Antwerp
  - 032-002_UCL Brussels, Brussels
  - 032-003_AZ Maria Middelares, Ghent
  - 032-001_University Hospital Brussel, Jette
  - Site 032-007_AZ Sint Maarten, Mechelen
- Spain (4):
  - 034-001_Hospital Clinic de Barcelona, Barcelona
  - 034-002_MD Anderson Cancer Center, Madrid
  - 034-003_Hospital Universitario Ramon y Cajal, Madrid
  - 034-004_Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: Undecided